CLINICAL TRIAL: NCT00197405
Title: Comparative Study of Fecal RNA Test With Immunochemical Fecal Occult Blood Test for Detecting Colorectal Cancer and Adenoma
Brief Title: Comparison of Fecal Ribonucleic Acid (RNA) Test With Fecal Occult Blood Test (FOBT) for Detecting Colorectal Cancer and Adenoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamamatsu University (Other)
Responsible Party: Shigeru Kanaoka, Hamamatsu University School of Medicine
Other Study IDs: CRC-FRT-001
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — freces, biopsy tissue samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Colorectal cancer (CRC) is the second common cause of death in the Western world, and is very increasing in Japan. Fecal occult blood test (FOBT) is used routinely for CRC screening, which has been shown to reduce the incidence, morbidity, and mortality of CRC. However, there is a need to develop a novel method to improve sensitivity. The investigators reported that Fecal COX-2 assay, one of fecal RNA test, is potentially useful for colorectal cancer screening (Gastroenterology 127; 422-427, 2004). So the investigators planed to compare fecal RNA test with FOBT for detecting colorectal cancer and adenoma.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of colorectal cancer or adenoma
* Subjects with no abnormal findings of colon

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: outpatients and inpatients of hospitals, subjects of parimary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 1999-08; Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Kanaoka, M.D., Study Chair
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Japan